CLINICAL TRIAL: NCT03783117
Title: Reducing Blood Viscosity and Suppressing Turbulence With Magneto-rheology to Lower Blood Pressure
Brief Title: Magneto-rheology to Lower Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardiovascular Therapy LLC (Industry)
Responsible Party: Principal Investigator, Rongjia Tao, Chief Scientist and Chief Counsel, Cardiovascular Therapy LLC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201801
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Subjects in second stage of hypertension: the systolic blood pressure in a range of 140-180 mmHg or diastolic blood pressure in a range 90-120 mmHg. For safety, subjects, who have a pacemaker or other metallic devices implanted, will not be admitted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Magnetic field treatment (Experimental): Each subject will place his/her right arm into a bore of the Magnetic Blood Pressure Lowering (MBPL) Device for magnetic treatment of 15 minutes, while the blood pressure is monitored with the left arm. The MBPL device produces a magnetic field around 1T parallel to the blood flow inside the arm. The subject's blood pressure will be lowered. The subject needs to come back to check the blood pressure 24 hours after the treatment.
  Interventions: Device: Magnetic field treatment

INTERVENTIONS:
Device: Magnetic field treatment — The MBPL device for clinical trials is made with modification of an electromagnet: A bore of 10cm diameter was made to go through the frame and poles. The device can produce a magnetic field close to 1.0 T inside the bore, which is along the axis direction. The trial for each subject takes about 20-30 minutes. To start with, the subject's blood pressure is measured first as the baseline. Afterwards, the subject places his/her right arm into the bore of the electromagnet for treatment while the blood pressure is monitored with the left arm. The magnetic treatment lasts about 15 minutes and will lower the subject's blood pressure. In order to see how long the effect lasts, the subject needs to return and measure the blood pressure again 24 hours after the treatment. The clinical trials are non-invasive. There is no medicine or surgery involved.

SUMMARY:
Heart attacks and strokes are the leading causes of death in US. High blood viscosity and turbulence in blood flow are the key for cardiovascular diseases. Recent research has shown that application of a strong magnetic field along the blood flow direction will polarize the red blood cells and align them into short chains along the flow, so that the blood viscosity in the flow direction is reduced significantly and disturbed motions in the directions perpendicular to the flow is suppressed. This makes the blood flow laminar, turbulence suppressed, and the possibility of cardiac events reduced. Such magnet treatment also cures rouleaux and improves the blood's oxygen function. The lab tests also confirm that the above effects last more than 24 hours after one treatment.

The purpose of this trial is to apply this technology to humans. According to the lab tests, this magnetic treatment has the potential to bring the following benefits to the subjects: (a)The blood viscosity will be reduced by 10-20% or more. (b) The turbulence in blood circulation will be suppressed by the treatment. After the treatment, the blood flow will be laminar. As a joint effect of viscosity reduction and turbulence suppression, the blood pressure will be lowered by 10-20% or more. (c) The subject's blood oxygen function will be improved by the treatment. Especially, if the subject has rouleaux in his/her blood, the effect will be significant. (d) The above effects will last for about 24 hours after one treatment and slowly decay; however, re-treatment will bring the effects back. (e) Because steady laminar blood flow is atheroprotective by active reduction of inflammatory genes, the magnetic treatment, reducing disturbed blood flow hemodynamics, would be possible to have a long term effect as an anti-atherogenic therapy if the treatment keeps for a while.

The investigators have just completed the pilot clinical trial. The tests confirm that the technology is safe and effective in lowering the blood pressure and the effect lasts about 24 hours. The present pivotal clinical trials are the continuation and expansion of the pilot tests. The successful clinical trials will make this technology available for people in preventing heart attack and stroke.

DETAILED DESCRIPTION:
GOAL: Conduct pivotal clinical trials with Magnetic Blood Pressure Lowering (MBPL) Device, developed in this lab, to see how effective it can lower patients' high blood pressure. The pilot study has confirmed the safety and performance of the device. The pivotal tests will test a large population of subject with hypertension to determine the effectiveness of the MBPL device and check if there is any adverse effect.

RECRUITMENT: For the pivotal clinical trials, subjects in second stage of hypertension will be selected: the systolic blood pressure in a range of 140-180 mmHg or diastolic blood pressure in a range 90-120 mmHg. For safety, subjects, who have a pacemaker or other metallic devices implanted, will not be selected. In addition, any adults unable to consent, cognitively impaired adults, and subjects who are not yet adults (infants, children, teenagers), pregnant women, and prisoners, will not be admitted.

STUDY: The MBPL device for clinical trials is made with modification of an electromagnet: A bore of 10 cm diameter was made to go through the frame and poles. The device can produce a magnetic field close to 1.0 T inside the bore, which is along the axis direction. The trial for each subject takes about 20-30 minutes. The subject's blood pressure will be measured first. Afterwards, the subject will place his/her right arm into the bore of the electromagnet for treatment while the blood pressure is monitored with the left arm. The magnetic treatment will last about 15 minutes.

In order to see how long the effect lasts, the subject needs to return and measure the blood pressure again 24 hours after the treatment. The clinical trials are non-invasive. There is no medicine or surgery involved.

ANALYSES: During the magnetic treatment, the MBPL device applies a strong magnetic field along the blood flow direction in subjects' right arm. Under the magnetic field, the deoxygenated red blood cells are polarized and form short chains along the blood flow direction. The blood circulation brings these chains to the whole body. Based on the lab results, the blood viscosity along the flow direction will be reduced by 10-20% or more; the turbulence in blood circulation will be suppressed by the treatment if the subject has turbulence in the blood circulation. As a result, the blood flow will become laminar and the blood pressure will be lowered. The above effects will last for about 24 hours after the treatment and slowly decay. However, re-treatment will bring the effects back. In long term, the magnetic treatment could prevent development of atherosclerotic plaques in blood vessels. The effectiveness of the magnetic treatment will be determined by

* evaluating the reduction of the systolic blood pressure and diastolic blood pressure immediately after the magnetic treatment;
* comparing the blood pressure 24 hours after the magnetic treatment with the initial blood pressure before the magnetic treatment and evaluating any reduction.

ELIGIBILITY:
Inclusion Criteria:

* The systolic blood pressure in a range of 140-180 mmHg or diastolic blood pressure in a range 90-120 mmHg.

Exclusion Criteria:

* Subjects with a pacemaker or other metallic devices implanted.
* Adults unable to consent,
* Cognitively impaired adults,
* Pregnant women,
* Prisoners.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-08-09 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Change of Blood Pressure at the End of Magnetic Treatment | Through study completion, an average of 1 year
  Measure and evaluate the change of both systolic blood pressure and diastolic blood pressure from the baseline at the end of magnetic treatment.

SECONDARY OUTCOMES:
Change of Blood Pressure 24 Hours after the Magnetic Treatment | Through study completion, an average of 1 year
  Measure and evaluate the change of both systolic blood pressure and diastolic blood pressure from the baseline 24 hours after the magnetic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rongjia Tao, Ph.D., Principal Investigator — Cardiovascular Therapy LLC
Locations (1):
- Magnetic Blood Pressure Lowering Device Study, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tao R, Huang K. Reducing blood viscosity with magnetic fields. Phys Rev E Stat Nonlin Soft Matter Phys. 2011 Jul;84(1 Pt 1):011905. doi: 10.1103/PhysRevE.84.011905. Epub 2011 Jul 12. PMID 21867211
- [Result] Tao R, Tang H, Xu X, Tawhid-Al-Islam K, Du E, "Systems and methods for reducing the viscosity of blood, suppressing turbulence in blood circulation, and curing rouleaux" PCT/US2017/059446, WO2018/085330A4
- See also: Special Report — http://www.aps.org/publications/apsnews/201705/magnetic.cfm
- Available data/document: Clinical Study Report — https://www.facebook.com/Cardiovasculartherapy/?modal=admin_todo_tour — After the clinical trials are completed, the clinical study report will be provided upon request via rtao@temple.edu.